CLINICAL TRIAL: NCT07344844
Title: Intérêt de la radiothérapie Adaptative en stéréotaxie Prostatique
Brief Title: Adaptive Stereotactic Radiotherapy for Localized Prostate Cancer
Acronym: SPAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Sainte Clotilde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A00339-40
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: SBRT; Cyberknife; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated by SBRT with pre-session low-dose CT (Other): Five low-dose, non-contrast CT scans performed immediately before each SBRT session (≈10 min before treatment) to assess anatomical variations impacting target volume and organ-at-risk dosimetry.
  Interventions: Other: Low-dose CT imaging before each SBRT session

INTERVENTIONS:
Other: Low-dose CT imaging before each SBRT session — Five low-dose, non-contrast CT scans performed immediately before each SBRT session (≈10 min before treatment) to assess anatomical variations impacting target volume and organ-at-risk dosimetry.

SUMMARY:
This study evaluates whether adaptive stereotactic body radiotherapy (SBRT) provides dosimetric advantages compared to non-adaptive SBRT in localized prostate cancer. Five low-dose CT scans are performed before each SBRT session to assess anatomical variations (bladder filling, rectal volume) and determine if a dosimetric recalculation would have been required. The study also evaluates cumulative dose to organs at risk, patient-reported quality of life over 24 months, and overall and recurrence-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Male aged ≥60 years
* Localized prostate cancer of low or intermediate risk (T1-T2)
* Gleason score 6-7
* PSA <15 ng/mL
* No evidence of metastatic disease
* Radiotherapy indicated for prostate cancer
* Affiliated with or benefiting from a French social security system
* French-speaking patient
* Patient appropriately informed and having signed a written informed consent form

Exclusion Criteria:

* Unable to read, write, or understand French
* Vulnerable patient as defined by Article L1121-6 of the French Public Health Code
* Adult under guardianship, curatorship, or legal protection ("sauvegarde de justice")
* Patient unable to personally provide informed consent according to Article L1121-8 of the French Public Health Code
* Patient already included in another interventional study that could interfere with study outcomes
* History of urological (prostate) or digestive surgery that could influence study outcomes
* Refusal to sign the written informed consent form

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring dosimetric recalculation due to anatomical variations | At each of the 5 SBRT sessions (10 days max) Based on scanners low-dose comparison.
  Percentage of patients for whom at least one stereotactic body radiotherapy (SBRT) fraction would have required a dosimetric recalculation due to anatomical variations (bladder filling and/or rectal emptying), based on comparison between the initial treatment plan and pre-treatment low-dose CT scans acquired before each SBRT fraction (5).
  This outcome reflects the potential benefit of an adaptive radiotherapy approach compared to a non-adaptive strategy.

SECONDARY OUTCOMES:
Cumulative delivered dose to Organs at Risk (OARs) | From baseline CT + all 5 fraction low-dose CT scans. (up to 10 days)
  Definition:
  Quantitative assessment of the dose actually delivered to each OAR across all fractions, based on dose-volume parameters derived from the low-dose CTs and DVH (Dose-Volume Histogram) analyses.
  OARs and parameters include:
  Rectum Maximum dose (0.03 cc) Dose to 3 cc Dose to 10%, 20%, and 50% of the volume
  Bladder Maximum dose (0.03 cc) Dose to 10% and 50% of the volume Penile bulb Maximum dose Dose to 3 cc
  Femoral heads Dose to 10 cc (combined left and right) Maximum dose
  Bowel (GETUG-14 constraints) D5cc D1cc
  Urethra Maximum dose
Change from baseline in global quality of life (EORTC QLQ-C30) | Time Frame: Baseline (pre-radiotherapy) 1 month 3 months 6 months 12 months 18 months 24 months post-radiotherapy
  Change from baseline in global quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
  Score range: 0-100 Higher scores indicate better quality of life.
Survival outcomes | 1, 3, 6, 12, 18, 24 months post-radiotherapy
  Overall Survival (OS): Death from any cause.
Recurrence-Free Survival (RFS) | 1, 3, 6, 12, 18, 24 months post-radiotherapy
  Clinical, biochemical, or radiological recurrence.
Change from baseline in prostate cancer-specific quality of life (EORTC QLQ-PR25) | Baseline, 1, 3, 6, 12, 18, and 24 months post-radiotherapy
  Change from baseline in prostate cancer-specific quality of life domains assessed using the EORTC QLQ-PR25 questionnaire.
  Score range: 0-100 Higher scores indicate worse symptoms.
Change from baseline in urinary symptoms (IPSS) | Baseline, 1, 3, 6, 12, 18, and 24 months post-radiotherapy
  Change from baseline in urinary symptoms assessed using the International Prostate Symptom Score (IPSS).
  Score range: 0-35 Higher scores indicate worse urinary symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Slama, Study Chair — Clinique Sainte Clotilde
Locations (1):
- Clinique Sainte Clotilde, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: Undecided